CLINICAL TRIAL: NCT02504476
Title: A Phase I, Randomized, Placebo-controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of AMG 581 in Healthy Subjects or Subjects With Schizophrenia or Schizoaffective Disorder on Antipsychotic Medication
Brief Title: Multiple Ascending Dose Study on Safety, Tolerability, and Pharmacokinetics of AMG 581 in Healthy Subjects or Subjects With Schizophrenia or Schizoaffective
Acronym: MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20130259
Record Dates: First submitted 2015-07-08; First posted 2015-07-22 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Schizophrenia or Schizoaffective Disorder
Keywords: Schizophrenia or Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- AMG 581 - Dose 1 (Active Comparator)
  Interventions: Drug: AMG 581
- AMG 581 - Dose 2 (Active Comparator)
  Interventions: Drug: AMG 581
- AMG 581 - Dose 3 (Active Comparator)
  Interventions: Drug: AMG 581
- AMG 581 - Dose 4 (Active Comparator)
  Interventions: Drug: AMG 581
- Placebo - Dose 1 (Placebo Comparator)
  Interventions: Drug: AMG 581; Drug: Placebo
- Placebo - Dose 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo - Dose 3 (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo - Dose 4 (Placebo Comparator)
  Interventions: Drug: Placebo
- AMG 581/Midazolam - Drug Interaction (Other)
  Interventions: Drug: AMG 581; Drug: Midazolam

INTERVENTIONS:
Drug: AMG 581 — Active drug
  Arms: AMG 581 - Dose 1; AMG 581 - Dose 2; AMG 581 - Dose 3; AMG 581 - Dose 4; AMG 581/Midazolam - Drug Interaction; Placebo - Dose 1
Drug: Placebo — Placebo
  Arms: Placebo - Dose 1; Placebo - Dose 2; Placebo - Dose 3; Placebo - Dose 4
Drug: Midazolam — Interaction
  Arms: AMG 581/Midazolam - Drug Interaction

SUMMARY:
The purpose of this study is to find out the time it takes to absorb, distribute, breakdown and remove the drug from the body in healthy participants and subjects with schizophrenia and whether it causes any side effects.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetic profile of ascending multiple oral doses of AMG 581 in healthy subjects or subjects with schizophrenia or schizoaffective disorder on antipsychotic medication. The study will also assess the effects of AMG 581 on midazolam PK in healthy subjects or subjects with schizophrenia or schizoaffective disorder on antipsychotic medication.

ELIGIBILITY:
Inclusion Criteria:

- Provided informed consent prior to initiation of any study-specific activities/procedures; -male or female subjects should be between the ages of 18 and 45 years (18-55 years for subjects with schizophrenia);-non-nicotine or non-tobacco (healthy subjects only); - no history of relevant medical disorders; - BMI ≥ 18.0; - females of non-reproductive potential; - males practicing effective birth control; - avoid tanning/direct sunlight; - schizophrenia or schizoaffective disorder; PANSS score ≤ 4 points on following items (i.e. conceptual disorganization, hallucinatory behavior, excitement, suspiciousness/persecution, hostility, depression, anxiety, disorientation, uncooperativeness, disturbance of volition, and poor impulse control) / total score ≤ 80 points

Exclusion Criteria:

* females lactating/breastfeeding; pregnant partners of male subjects; essential tremor or gait disturbance; - history of hereditary shorten QT syndrome; - malignancy or tumor (other than skin cancers); - history of GI disease that could interfere with absorption; - QTc ≥ 450 msec or ≤ 380 msec; - HbA1c ≥ 7%;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Reported treatment-emergent adverse events | 39 days
  Number and percent of subjects experiencing adverse events
Changes in systolic/diastolic blood pressure | 39 days
  Summaries over time and/or changes from baseline over time in systolic and/or diastolic blood pressure
Changes in heart rate | 39 days
  Summaries over time and/or changes from baseline over time in heart rate
Changes in respiratory rate | 39 days
  Summaries over time and/or changes from baseline over time in respiratory rate
Changes in temperature | 39 days
  Summaries over time and/or changes from baseline over time in temperature
Changes in ECGs | 39 days
  Summaries over time and/or changes from baseline over time in ECGs
Maximum change from baseline in QTc in ECGs and number and percentage of subjects with maximum changes exceeding prespecified limits in each group | 39 days
  Subjects' maximum change from baseline in QTc and the number and percentage of subjects in each group
Maximum post-baseline QTc values and number and percentage of subjects with maximum post-baseline QTc values exceeding prespecified limits in each group | 39 days
  Subjects' maximum post-baseline values and the number and percentage of subjects in each group
Scores at each study visit for Simpson Angus Scale (SAS) | 39 days
  Summaries over time and/or changes from baseline over time in changes in Simpson Angus Scale (SAS) score
Scores at each study visit for Barnes Akathisia Rating Scale (BARS) | 39 days
  Summaries over time and/or changes from baseline over time in in Barnes Akathisia Rating Scale (BARS) score
Subject incidence of treatment-emergent suicidal ideation and behavior as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) | 39 days
  Subject incidence of treatment-emergent suicidal ideation and behavior as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) summarized by cohort

SECONDARY OUTCOMES:
Compare PK parameter (Cmax) between Day 1 and Day 18 | 18 days
  Compare PK parameter (Cmax) between Day 1 and Day 18
Compare PK parameter (AUC) between Day 1 and Day 18 | 18 days
  Compare PK parameter (AUC) between Day 1 and Day 18
Compare PK parameter (tmax) Compare PK parameter (tmax) between Day 1 and Day 18 | 18 days
  Compare PK parameter (tmax) Compare PK parameter (tmax) between Day 1 and Day 18
Plasma PK parameters of midazolam and 1-OH midazolam | 36 days
  Cmax and AUC prior to versus following AMG 581 administration

OTHER OUTCOMES:
AMG 581 metabolites in plasma | 39 days
  Metabolites of AMG 581 in plasma
Cmax and AUC of AMG 581 prior to versus following midazolam administration | 36 days
  Cmax and AUC prior to versus following AMG 581 administration
Subjective experience following administration of AMG 581 | 39 days
  Subjective experience of study subjects following administration of AMG 581 as measured by the Bond and Lader visual analogue scales (VAS)
Changes in psychotic symptoms following administration of AMG 581 | 39 days
  Subjective experience of study subjects following administration of AMG 581 as measured by the Positive and Negative Syndrome Scale (PANSS) (subjects with schizophrenia or schizoaffective disorder receiving antipsychotic treatment only)
Relationship between QTc and temperature | 39 days
  To explore the relationship between changes in QTc and changes in body temperature

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- United States (2):
  - Research Site, Glendale, California
  - Parexel, Glendale, California

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com